CLINICAL TRIAL: NCT03916900
Title: Evaluation of Postoperative Pain and Success Rate After Pulpotomy Versus Root Canal Treatment in Cariously Exposed Mature Permanent Molars: A Randomized Controlled Trial
Brief Title: Postoperative Pain and Success Rate in Pulpotomy Versus Root Canal Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Aya Alaa Abdelaziz Elsayed, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 14422017490583
Record Dates: First submitted 2019-04-11; First posted 2019-04-16 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Pulpitis - Irreversible
Keywords: Pulpotomy; Root canal treatment; Mature; Cariously exposed; Permanent molars; Irreversible pulpitis
MeSH Terms: interventions — Pulpotomy

STUDY DESIGN:
Intervention Model Description: Parallel assignment
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pulpotomy (Experimental): Group A (Experimental group) Pulpotomy:
  The teeth will be anesthetized with 4% articaine 1:100,000 epinephrine (Artinibsa®; Inibsa Dental, Lliçà de Vall, Spain) by inferior alveolar nerve block.Under rubber dam isolation, pulpotomy will be performed with a large sterile round end bur in a high speed hand piece with copious irrigation; pulp tissue will be removed by a sharp spoon excavator to the orifice level. Hemostasis will be achieved by the application of a wet cotton pellet moistened with 2.5% NaOCL for 2 min and repeated if needed.
  After hemostasis, Biodentine (Septodont, Saint Maur des Fausses, France) will be mixed according to the manufacturer's instructions and gently placed over the pulp to thickness of 2-3 mm.Biodentine will be covered by resin modified glass-ionomer and teeth will be restored using composite resin.A postoperative radiograph will be taken by parallel technique.
  Interventions: Procedure: Pulpotomy
- Root canal treatment (Active Comparator): Group B (control group) Root canal treatment:
  The teeth were anesthetized with 4% articaine 1:100,000 epinephrine (Artinibsa®; Inibsa Dental, Lliçà de Vall, Spain).Under rubber dam isolation, root canal treatment will be performed in single visit.Working length will be determined using stainless steel k-files (Mani, Inc.) keeping 0.5 to 1.0 mm short of the apex using a RootZX apex locator (J. Morita, Irvine, CA) and confirmed radiographically. Mechanical preparation will be achieved by a crown-down technique using using the M-PRO system (IMD, Shanghai, China) and irrigation with 5 mL 2.5% NaOCl between instruments.Obturation will be done with gutta-percha (Meta Biomed Co. Ltd, Cheongwongun, Chungbuk, Korea) and resin sealer ADseal (Meta Biomed CO., LTD, Korea) using cold lateral condensation technique and restored with composite resin with a base of glass-ionomer cement. A postoperative radiograph will be taken by parallel technique.
  Interventions: Procedure: Root canal treatment

INTERVENTIONS:
Procedure: Pulpotomy — Pulpotomy is a procedure in which the coronal pulp is amputated, and the remaining radicular pulp tissue is treated with a medicament to preserve the pulp's health .This technique involves administration of local analgesia, Isolation of the tooth with rubber dam, Complete caries removal and then access to the pulp chamber using drills
  Arms: Pulpotomy
Procedure: Root canal treatment — Root canal treatment is an often straightforward procedure to relieve dental pain and save teeth. Patients typically need a root canal when there is inflammation or infection in the roots of a tooth. During root canal treatment, an endodontist who specializes in such treatment carefully removes the pulp inside the tooth, cleans, disinfects and shapes the root canals, and places a filling to seal the space.
  Arms: Root canal treatment

SUMMARY:
Pulpotomy has been proposed in the last decade as a definitive treatment of mature permanent teeth with irreversible pulpitis due to the better understanding of the pulp biology and development of bioactive materials . This technique involves removal of the coronal portion of the pulp that has undergo degenerative and irreversible changes to the level of the canal orifices and leaving the healthy vital radicular portion of the pulp. The surrogate marker for the degree of inflammation and the healing potential of the remaining pulp tissue has been suggested to be the ability to control the bleeding after pulp amputation.

By preserving the pulp vitality, this can help in maintaining proprioceptive, reparative, innervation (tooth sensitivity), vascularization, and damping functions. The vital pulp can continue to serve the function of protecting the tooth from overload by means of protective feedback mechanism and preventing fracture because of the presence of pulp and organic tissue in the dentinal tubules..

DETAILED DESCRIPTION:
The routine dental treatment for the patient diagnosed with symptomatic or asymptomatic irreversible pulpitis secondary to deep carious lesion is conventional root canal treatment. Root canal treatment is the preferred treatment option because of its superior success rate to other treatments .

However, it is expensive, time consuming and complicated. Root canal treatment needs special clinical skills and high socio-economic status to afford the cost of the treatment. Unfortunately, in developing countries these can be un-reachable. Therefore, extraction is the only alternative option to the affected teeth . Moreover, a recent systematic review by Ng et al stated that the success rate of root canal treatment had not improved over the past few decades and molars had poor survival rates in comparison to non-molar teeth.In addition, It was stated that the survival rate of endodontically treated tooth is alarmingly low in comparison to vital teeth, especially molars, During root canal treatment many mishaps can occur such as perforations, ledges and extrusion of root filling, that reduces the longevity of root treated teeth .

Carious pulp exposure of permanent molars in children is a very common unfortunate event faced in Pediatric Dentistry and Public Health department in Cairo university. This may be due to the low socioeconomic status, ignorance of patients attending that clinic, their wrong eating habits and their bad oral hygiene.

Root canal treatment in an uncooperative young patient is very complicated which may affect the quality and prognosis of the treatment itself. Therefore, an economical, simple and conservative technique such as pulpotomy should be considered Pulpotomy has been proposed in the last decade as a definitive treatment of mature permanent teeth with irreversible pulpitis due to the better understanding of the pulp biology and development of bioactive materials . This technique involves removal of the coronal portion of the pulp that has undergo degenerative and irreversible changes to the level of the canal orifices and leaving the healthy vital radicular portion of the pulp. The surrogate marker for the degree of inflammation and the healing potential of the remaining pulp tissue has been suggested to be the ability to control the bleeding after pulp amputation..

By preserving the pulp vitality, this can help in maintaining proprioceptive, reparative, innervation (tooth sensitivity), vascularization, and damping functions.The vital pulp can continue to serve the function of protecting the tooth from overload by means of protective feedback mechanism and preventing fracture because of the presence of pulp and organic tissue in the dentinal tubules.The dentin -pulp complex will stimulate the formation of tertiary dentine or a mineralized barrier protecting itself .

Compared to the root canal treatment, pulpotomy is considered less technique sensitive so it can be performed by general dental practitioners. Hence, It increases the patients' access to dental care and more clinicians will be able to provide the affordable treatment saving more teeth when the patients cannot afford the root canal treatment leaving extraction as a last treatment option.

It is believed that the pulp tissue of the younger aged patients has higher healing capacity and regenerative powers than pulp tissue in older aged patients.

ELIGIBILITY:
Inclusion Criteria:

* Children from 9 to 15 years, in good general health and medically free.
* Cariously exposed mature (complete root formation length and apical closure) permanent molars with reversible pulpitis, symptomatic or asymptomatic irreversible pulpits.
* Teeth should be vital on cold testing.
* Restorable teeth.
* Vital bleeding present in all canals.
* Hemostasis achieved after complete pulpotomy.
* Preoperative radiograph:Absence of periapical or inter-radicular radiolucency, widening of PDL space, internal or external root resorption.

Exclusion Criteria:

* Children with systemic diseases physical or mental disability, unable to attend follow-up visits or refuse participation.
* Previously accessed teeth.
* Necrotic teeth (negative response to cold testing or absence of bleeding after access cavity).
* Presence of sinus tract or swelling.
* Excessive bleeding after pulpotomy and not controlled after several minutes.
* Teeth with marginal periodontitis or crestal bone loss.

Ages: 9 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 52 (Estimated)
Dates: Start 2019-06-01 (Estimated); Primary Completion 2020-06-01 (Estimated); Study Completion 2020-07-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain: VAS (visual analogue scale) | 4 days postoperatively
  Postoperative pain reported by the patient after pulpotomy and root canal treatment by VAS (visual analogue scale).Scale from 0-10 recorded every 24hours until the fourth day. The VAS for pain is a straight line with one end (point 0) meaning no pain and the other end( point 10) meaning the worst pain imaginable

SECONDARY OUTCOMES:
Swelling, sinus or fistula | 9 months
  They will be assessed by visual examination.(Binary)
Pain on percussion | 9 months
  It will be assessed by percussion test .(Binary)
Radiographic success | 9 months
  It is defined as absence of inter-radicular or periapical radiolucency, widening of PDL space, internal or external root resorption).It will be assessed by periapical radiograph. parallel technique. Interpretation by Cohen's Kappa will be calculated.

IPD SHARING:
Plan to Share IPD: Yes
study protocol, informed consent, clinical study report
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 9 months after completion of the study
Access Criteria: ClinicalTrials.gov
URL: http://ClinicalTrials.gov